CLINICAL TRIAL: NCT06923852
Title: Acute Respiratory Disease as a Fulcrum Point to Quit Smoking: Evaluation of an ED-based Intervention
Acronym: Intervention
Status: Completed | Type: Observational
Sponsor: Seda Oğuz (Other)
Responsible Party: Sponsor-Investigator, Seda Oğuz, Emergency Physician, Haydarpasa Numune Training and Research Hospital
Organization: Haydarpasa Numune Training and Research Hospital (Other)
Other Study IDs: SMOKE-21041991
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Emergency Department Visit; Acute Respiratory Infections (ARIs)
MeSH Terms: conditions — Smoking Cessation | interventions — World Health Organization; corticosteroid hormone-induced factor; Insemination, Artificial, Heterologous

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Active smokers who attend the emergency depertment with acute respiratory infections
  Interventions: Behavioral: Smoking cessation support that World Health Organization (WHO) 5A model (Ask, Advise, Assess, Assist, Arrange).

INTERVENTIONS:
Behavioral: Smoking cessation support that World Health Organization (WHO) 5A model (Ask, Advise, Assess, Assist, Arrange). — Smoking cessation support that World Health Organization (WHO) 5A model (Ask, Advise, Assess, Assist, Arrange).

SUMMARY:
This study aims to evaluate smoking cessation success rates using the Fagerström Test for Nicotine Dependence (FTND) in smoking cessation treatment. The study has a retrospective design, analyzing data from patients who applied to a smoking cessation clinic to investigate the impact of nicotine dependence severity on quitting success.

DETAILED DESCRIPTION:
Emergency departments (EDs) are among the most critical referral centers for individuals with health problems resulting from the direct and indirect effects of smoking. Individuals may be more motivated to change their smoking habits, especially during acute attacks of respiratory diseases. The American College of Emergency Physicians (ACEP) and some organizations recommend that interventions for smoking cessation should be implemented by physicians and nurses in the form of counseling for patients with active smoking who receive treatment for acute respiratory infections (ARI) in EDs. However, interventions for smoking cessation are frequently performed in primary health care institutions and according to studies, a high majority of emergency physicians think that EDs are not the appropriate place for this intervention and are not included in their professional responsibilities.

The effect of nicotine dependence (ND) severity on smoking cessation has been shown in studies. Fagerström Test of Nicotine Dependence (FTND) developed by Fagerström et al. is a widely used tool to measure the ND level of individuals. The Turkish validity and reliability study of the test was conducted by Uysal et al. In the approach to smoking cessation, ND level comes to the forefront in determining personalized intervention strategies. At high levels of addiction, nicotine replacement therapy or pharmacologic support is recommended because the physical and psychological dependence of individuals is more intense. In these cases, motivational counseling and regular follow-up are necessary during the cessation process. At moderate levels of addiction, nicotine replacement products or behavioral therapies are usually recommended, while less pharmacological intervention may be required. At low levels of addiction, behavioral support and counseling may be sufficient for smoking cessation. Pharmacologic treatment is usually not needed in these individuals, but education and awareness-raising methods that support smoking cessation can be used. Intervention with strategies appropriate to the level of ND is a crucial factor in increasing the success of smoking cessation.

When determining the assistance method in individuals who want to quit smoking; WHO recommends five major steps (5A) in smoking cessation treatment. In practice, the "Ask, Advise, Assess, Assist, Arrange" approach is an evidence-based smoking cessation model that has been developed to provide effective interventions in a short time, especially in busy working environments.

This study aimed to examine the effects of short structured interviews with patients who presented to the ED due to ARI on smoking cessation behavior and to follow up for one month. It is aimed to evaluate the applicability of smoking cessation interventions on those with ARI in EDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were active smokers and admitted to the emergency department with acute respiratory system complaints.

Exclusion Criteria:

* Exclusion criteria included individuals under 18 years of age, ASA class III-IV, pregnancy or breastfeeding, communication difficulties such as language barrier or cognitive impairment, psychotic behaviors or history of psychiatric treatment, and initiation of smoking cessation treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20,928 patients presented to the ED during the specified period and 2,018 of these patients were evaluated with acute respiratory complaints diagnosed with ARI. Of the patients admitted with ARI, 541 reported active smoking. Finally, 288 participants were accepted for the study.
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-01-10 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Smoking cessation success on acute respiratory infections patients based on FTND score | Two periods as first week after intervention and first month after intervention.
  Examine the effects of short structured interviews with patients who presented to the ED due to ARI on smoking cessation behavior. It is aimed to evaluate the applicability of smoking cessation interventions on those with ARI in EDs.

IPD SHARING:
Plan to Share IPD: Undecided